CLINICAL TRIAL: NCT05245708
Title: The Modulatory Effects of Oxytocin on Reinforcement Learning and Interoceptive Processing
Brief Title: Effects of Oxytocin on Reinforcement Learning and Interoception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-83
Record Dates: First submitted 2022-02-07; First posted 2022-02-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: oxytocin; learning; interoception

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): a single dose of 24 international units (IU) of OT will be administered with 3 puffs of treatment to each nostril.
  Interventions: Drug: Intranasal oxytocin
- placebo (Experimental): a single dose of 24 international units (IU) of placebo will be administered with 3 puffs of treatment to each nostril.
  Interventions: Drug: intranasal placebo

INTERVENTIONS:
Drug: Intranasal oxytocin — Each subject will be assigned to intranasal administration of oxytocin (24 IU).
  Arms: oxytocin
Drug: intranasal placebo — Each subject will be assigned to intranasal placebo.
  Arms: placebo

SUMMARY:
The main aim of the study is to investigate whether intranasal oxytocin has effects on reinforcement learning under dynamic environment and interoceptive processing based on behavioral and electroencephalogram (EEG) responses.

DETAILED DESCRIPTION:
A double-blinded, placebo-controled, between-subject design is employed in this study. In a randomized order, a total of 80 healthy males are instructed to self-administrated intranasal spray of oxytocin or placebo. (1) Participants first complete a probabilistic reward learning task 45 minutes after treatment with behavioral (response time and accuracy) and EEG data (ERP components such as FRN, ERN and P300) being collected during this task. (2) A resting-state recording and a heartbeat counting task are conducted following the learning task with ECG and EEG data being collected. Personality traits of subjects are assessed using validated Chinese version questionnaires including the Beck Depression Inventory (BDI-II), State-Trait Anxiety Inventory (STAI), Autism Spectrum Quotient (ASQ), the Cognitive Flexibility Inventory(CFI), Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ), Behavioral Inhibition System and Behavioral Activation System Scale (BIS/BAS). Subjects are asked to complete Positive and Negative Affect Schedule (PANAS) when they just arrive, before and after the tasks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders.

Exclusion Criteria:

* History of brain injury medical or mental illness.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Behavioral index in the learning task: chioce accuracy | 45-65 minutes after treatment administration
  The accuracy of subjects choosing the better option.
Behavioral index in the heartbeat counting task: interoceptive accuracy | 65-75 minutes after treatment administration
  Individuals' ability to perceive internal cardiac signals

SECONDARY OUTCOMES:
ERP components in the learning task: ERN, FRN, P300, N2pc | 45-65 minutes after treatment administration
  ERN and FRN are indices of reward expectancy and prediction error in reinforcement learning. P300 is associated with attention allocation. N2pc is an early component associated with visual selective attention.
ERP components in the heartbeat counting task: heartbeat-evoked potential (HEP) | 65-75 minutes after treatment administration
  HEP is a scalp event-related potential that reflects cortical processing of cardiac interoceptive signals

CONTACTS AND LOCATIONS:
Overall Officials: Yao Shuxia, Dr, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China (UESTC), Chengdu, Sichuan, China